CLINICAL TRIAL: NCT01010997
Title: Foresee Home for Monitoring Age Related Macular Degeneration (AMD)
Acronym: Foresee Home
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Sponsor
Organization: Notal Vision Inc. (Industry)
Other Study IDs: FORESEE HOME- 02; 75909 (Other: Local IRB)
Record Dates: First submitted 2009-11-08; First posted 2009-11-10 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD, CNV
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Dry AMD: Intermediate AMD subjects
  Interventions: Device: Foresee Home
- Wet - treated AMD: AMD subjects under treatments
  Interventions: Device: Foresee Home

INTERVENTIONS:
Device: Foresee Home — using the Foresee home device

SUMMARY:
The FORESEE HOME is intended for the early detection of central and paracentral irregularities (abnormalities) in the visual field, most commonly associated with AMD. However, the device has ability to detect the development of the lesion post treatment and therefore to asses in determination of the next treatment.

DETAILED DESCRIPTION:
The FORESEE HOME is intended for the early detection of central and paracentral irregularities (abnormalities) in the visual field, most commonly associated with AMD. However, the device has ability to detect the development of the lesion post treatment and therefore to asses in determination of the next treatment.

The OCT May be use as well to identify choroidal neovascularization (CNV). Comparison between the two methods will allow better understanding of both devices.

The FORESEE HOME can use as an assessment tool for the progression and success of the treatment given to AMD lesions. Therefore, evaluation the size and the location of the treated lesions may serve as an additional tool.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study
* Subjects diagnosed as CNV under treatment or Intermediate AMD in at least one eye
* Did not perform more then 10 anti- VEGF injections
* Age >50 years
* VA with habitual correction >6/45 in the study eye
* Computer users

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy,
* Any non-macular related ocular surgery performed within 3 months prior to study entry in the target eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AMD subjects
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To investigate the FORESEE HOME ability to diagnose AMD in different stages | 1 year

SECONDARY OUTCOMES:
To investigate the correlation between visual fields (VF) defects map generated by the FORESEE HOME and features of the choroidal neovascular lesions (CNV) demonstrated by Optical Coherence Tomography(OCT). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eliezer Kraus, MD, Principal Investigator — Naharia Hospital
Locations (1):
- Naharia Hospital, Nahariya, Israel